CLINICAL TRIAL: NCT02299570
Title: A Phase 2B Prospective, Randomized, Double-blinded, Placebo-controlled Clinical Study Demonstrating the Efficacy and Safety of Rebiotix RBX2660 (Microbiota Suspension) for the Treatment of Recurrent Clostridium Difficile Infection
Brief Title: Microbiota Restoration Therapy for Recurrent Clostridium Difficile Infection
Acronym: PUNCHCD2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rebiotix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-01
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Enterocolitis Clostridium Difficile Recurrent
Keywords: Clostridium difficile; C diff; CDI; CDAD; Fecal transplant; Fecal Microbiota Transplant; Diarrhea; FMT; Microbiota restoration therapy; Microbiota suspension; Fecal bacteriotherapy; C diff diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Active Comparator): Two enemas of RBX2660 (microbiota suspension) administered 7 days apart
  Interventions: Biological: RBX2660 (microbiota suspension)
- Group B (Placebo Comparator): Two enemas of placebo administered 7 days apart
  Interventions: Other: Placebo
- Group C (Active Comparator): 1 enema of RBX2660 (microbiota suspension) and 1 enema of placebo administered 7 days apart
  Interventions: Biological: RBX2660 (microbiota suspension); Other: Placebo

INTERVENTIONS:
Biological: RBX2660 (microbiota suspension) — A suspension of intestinal microbes
  Arms: Group A; Group C
Other: Placebo — A suspension of saline and cryoprotectant
  Arms: Group B; Group C

SUMMARY:
This is the first prospective, multi-center, double-blinded, randomized controlled study of a microbiota suspension derived from intestinal microbes. Patients who have had at least two recurrences of C. difficile infection (CDI) after a primary episode and have completed at least two rounds of standard-of-care oral antibiotic therapy or have had at least two episodes of severe CDI resulting in hospitalization may be eligible for the study. Patients whose CDI returns in less than 8 weeks after the last assigned study treatment may be eligible to receive up to 2 treatments with RBX2660 in the open-label portion of the study.

DETAILED DESCRIPTION:
This is the first prospective, multi-center, double-blinded, randomized controlled study of a microbiota suspension derived from intestinal microbes. The primary assessments for this study are (i) efficacy of RBX2660 compared to placebo at 8 weeks and (ii) safety via assessment of adverse events. Study visits are at 1-, 4- and 8-weeks after treatment with additional follow-up at 3, 6 12 and 24 months post treatment. Patients who have had at least two recurrences of C. difficile infection (CDI) after a primary episode and have completed at least two rounds of standard-of-care oral antibiotic therapy or have had at least two episodes of severe CDI resulting in hospitalization may be eligible for the study. Patients whose CDI returns in less than 8 weeks after the last assigned study treatment may be eligible to receive up to 2 treatments with RBX2660 in the open-label portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Medical record documentation of recurrent CDI either: a) at least two recurrences after a primary episode and has completed at least two rounds of standard-of-care oral antibiotic therapy or b) has had at least two episodes of severe CDI resulting in hospitalization.
* Documented history that the subject's recurrent CDI is controlled while on antibiotics even if the subject is not currently on antibiotics.
* A positive stool test for the presence of C. difficile within 60 days prior to enrollment.

Exclusion Criteria:

* A known history of continued C. difficile diarrhea while taking on a course of antibiotics prescribed for CDI treatment.
* Requires antibiotic therapy for a condition other than recurrent CDI.
* Previous fecal transplant prior to study enrollment.
* History of inflammatory bowel disease (IBD), e.g., ulcerative colitis, Crohn's disease, or microscopic colitis.
* History of irritable bowel syndrome (IBS).
* History of chronic diarrhea.
* History of celiac disease.
* Colostomy.
* Planned surgery requiring perioperative antibiotics within 6 months of study enrollment.
* Life expectancy of < 12 months.
* Compromised immune system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teena Chopra, MD MPH, Study Chair — Wayne State University
Locations (21):
- United States (19):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Colorado, Aurora, Colorado
  - Borland-Groover Clinic, Jacksonville, Florida
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Loyola University Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Infectious Diseases of Indiana, Indianapolis, Indiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New York Hospital Queens, Flushing, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical College, New York, New York
  - Gastroenterology Group of Rochester, Rochester, New York
  - Sanford Health, Fargo, North Dakota
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - Regional Infectious Diseases and Infusion Center, Lima, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - St. Joseph's Hospital, Hamilton, Ontario

REFERENCES:
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Moayyedi P, Marshall JK, Yuan Y, Hunt R. Canadian Association of Gastroenterology position statement: fecal microbiota transplant therapy. Can J Gastroenterol Hepatol. 2014 Feb;28(2):66-8. doi: 10.1155/2014/346590. No abstract available. PMID 25232572
- [Background] Gough E, Shaikh H, Manges AR. Systematic review of intestinal microbiota transplantation (fecal bacteriotherapy) for recurrent Clostridium difficile infection. Clin Infect Dis. 2011 Nov;53(10):994-1002. doi: 10.1093/cid/cir632. PMID 22002980
- [Derived] Lee C, Feuerstadt P, Louie T, Bancke L, Guthmueller B, Harvey A, Hoeyer F, Orenstein R, Dubberke ER, Khanna S. Integrated analysis of the safety of fecal microbiota, live-jslm in adults with recurrent Clostridioides difficile infection from five prospective clinical trials: an update. Therap Adv Gastroenterol. 2025 Nov 12;18:17562848251395566. doi: 10.1177/17562848251395566. eCollection 2025. PMID 41245385
- [Derived] Dubberke ER, Orenstein R, Khanna S, Guthmueller B, Lee C. Final Results from a Phase 2b Randomized, Placebo-Controlled Clinical Trial of RBX2660: A Microbiota-Based Drug for the Prevention of Recurrent Clostridioides difficile Infection. Infect Dis Ther. 2023 Feb;12(2):703-709. doi: 10.1007/s40121-022-00744-3. Epub 2022 Dec 21. PMID 36544075
- [Derived] Kwak S, Choi J, Hink T, Reske KA, Blount K, Jones C, Bost MH, Sun X, Burnham CD, Dubberke ER, Dantas G; CDC Prevention Epicenter Program. Impact of investigational microbiota therapeutic RBX2660 on the gut microbiome and resistome revealed by a placebo-controlled clinical trial. Microbiome. 2020 Aug 31;8(1):125. doi: 10.1186/s40168-020-00907-9. PMID 32862830
- [Derived] Dubberke ER, Lee CH, Orenstein R, Khanna S, Hecht G, Gerding DN. Results From a Randomized, Placebo-Controlled Clinical Trial of a RBX2660-A Microbiota-Based Drug for the Prevention of Recurrent Clostridium difficile Infection. Clin Infect Dis. 2018 Sep 28;67(8):1198-1204. doi: 10.1093/cid/ciy259. PMID 29617739
- See also: Sponsor website — http://www.rebiotix.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 12/10/14 to 11/13/15 at 21 medical clinics in the United States and Canada. Recruiment was performed by trained investigators and study coordinators.
Pre-assignment Details: Seventeen enrolled subjects did not proceed to randomization and were exited from the study. Of the 133 randomized subjects remaining, five subjects chose to withdraw prior to treatment and in one subject the first blinded enema was not able to be initiated due to anxiety and the subject subsequently chose to withdraw.
Groups:
- Group A: Two enemas of RBX2660 administered 7 days apart
  RBX2660 (microbiota suspension): A suspension of intestinal microbes
- Group C: 1 enema of RBX2660 and 1 enema of placebo administered 7 days apart
  RBX2660 (microbiota suspension): A suspension of intestinal microbes
  Placebo: A suspension of saline and cryoprotectant
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 45 | 44 | 44
Completed | 31 | 35 | 25
Not Completed | 14 | 9 | 19

BASELINE CHARACTERISTICS:
Population: This analysis population corresponds to the Intent to Treat Analysis Population. It includes subjects that were randomized into the treatment groups, but not treated, as well as one subject who was randomized into Group C, but received treatment as if in Group A.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 45 | 44 | 44 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 19 | 25 | 25 | 69
  >=65 years | 26 | 19 | 18 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (19.15) | 58.8 (19.24) | 61.0 (19.69) | 61.1 (19.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 25 | 81
  Male | 19 | 14 | 19 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 43 | 42 | 42 | 127
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 44 | 43 | 42 | 129
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 8 | 8 | 28
  United States | 33 | 36 | 36 | 105

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success of Group A (2 Doses of RBX2660) vs Group B (2 Doses of Placebo) (ITT)
Description: The primary endpoint is to evaluate treatment success, defined as the absence of CDAD without the need for retreatment with C. difficile anti-infective therapy or fecal transplant (FT) at 56 days after administration of the last assigned study enema, of Group A (two enemas of RBX2660) vs. Group B (two enemas of placebo).
Time Frame: 8 weeks after last assigned study treatment
Population: ITT - Subjects in the ITT that were randomized, but not treated, as well as subjects with an "indeterminate" treatment outcome, were also conservatively treated as treatment failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 45 | 44
Participants
  Treatment Success | 25 | 19
  Treatment Failure | 20 | 25

2. Secondary Outcome: Treatment Success Between Group C (1 Enema of RBX2660 and 1 Enema of Placebo) vs Group B (Two Enemas of Placebo) (ITT)
Description: Treatment Success was defined as the absence of CDAD without the need for retreatment with C. difficile anti-infective therapy or fecal transplant (FT) at 56 days after administration of the last assigned study enema
Time Frame: 8-weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Group B | Group C
Number analyzed (Participants) | 44 | 44
Participants
  Success | 19 | 25
  Failure | 25 | 19

3. Secondary Outcome: Treatment Success Evaluated Between Group A (Two Enemas of RBX2660) Versus Group C (1 Enema of RBX2660 and 1 Enema of Placebo) (ITT)
Description: Treatment success, defined as the absence of CDAD without the need for retreatment with C. difficile anti-infective therapy or fecal transplant (FT) at 56 days after administration of the last assigned study enema.
Time Frame: 8-weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group C
Number analyzed (Participants) | 45 | 44
Participants
  Success | 25 | 25
  Failure | 20 | 19

4. Secondary Outcome: SF-36 Scores Obtained at the 1-week, 4-week, and 8-week Assessments Visits During the Double-blind Period as Compared to Baseline (ITT)
Description: The validated SF-36 scale was used to identify changes to quality of life (QoL) following study treatment. Each component is analyzed on a norm-based scoring (0-100) with a higher score representing an improvement in QoL.
Time Frame: 8-week
Population: ITT
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 45 | 44 | 44
Score on a scale
  Physical Comp Baseline: number analyzed (Participants) | 39 | 44 | 42
  Physical Comp Baseline | 39.4 (11.4) | 39.4 (9.7) | 43.4 (10.5)
  Physical Comp Week 1: number analyzed (Participants) | 32 | 30 | 28
  Physical Comp Week 1 | 44.3 (10.2) | 45.0 (9.7) | 46.4 (10.1)
  Physical Comp Week 4: number analyzed (Participants) | 33 | 31 | 29
  Physical Comp Week 4 | 44.9 (11.6) | 45.6 (10.2) | 46.1 (11.2)
  Physical Comp Week 8: number analyzed (Participants) | 33 | 31 | 32
  Physical Comp Week 8 | 43.9 (10.9) | 45.8 (10.6) | 46.5 (12.1)
  Mental Comp Baseline: number analyzed (Participants) | 40 | 44 | 42
  Mental Comp Baseline | 44.6 (13.5) | 42.5 (11.5) | 45.0 (11.9)
  Mental Comp Week 1: number analyzed (Participants) | 32 | 30 | 28
  Mental Comp Week 1 | 51.8 (10.5) | 51.2 (10.3) | 50.6 (8.2)
  Mental Comp Week 4: number analyzed (Participants) | 33 | 31 | 29
  Mental Comp Week 4 | 53.5 (10.7) | 48.2 (12.4) | 51.5 (6.4)
  Mental Comp Week 8: number analyzed (Participants) | 33 | 31 | 32
  Mental Comp Week 8 | 52.1 (10.8) | 49.8 (11.7) | 51.2 (7.6)

5. Secondary Outcome: Time to CDAD Recurrence After Completion of the Assigned Study Treatment for Group A vs. Group B (ITT)
Description: Time to CDI Recurrence was evaluated using Kaplan-Meier Analysis and expressed by percentage of subjects who were recurrence free at a certain time point (every 7 days) from completion of the last blinded enema.
Time Frame: 8-weeks
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 45 | 44
percentage of participants
  % Recurrence Free by Day 0 | 91.1 | 100
  % Recurrence Free by Day 7: number analyzed (Participants) | 35 | 35
  % Recurrence Free by Day 7 | 73.3 | 77.3
  % Recurrence Free by Day 14: number analyzed (Participants) | 30 | 30
  % Recurrence Free by Day 14 | 66.7 | 63.6
  % Recurrence Free by Day 21: number analyzed (Participants) | 27 | 27
  % Recurrence Free by Day 21 | 60.0 | 61.4
  % Recurrence Free by Day 28: number analyzed (Participants) | 27 | 25
  % Recurrence Free by Day 28 | 60.0 | 56.8
  % Recurrence Free by Day 35: number analyzed (Participants) | 27 | 23
  % Recurrence Free by Day 35 | 57.8 | 52.3
  % Recurrence Free by Day 42: number analyzed (Participants) | 26 | 22
  % Recurrence Free by Day 42 | 57.8 | 50.0
  % Recurrence Free by Day 49: number analyzed (Participants) | 24 | 21
  % Recurrence Free by Day 49 | 55.5 | 47.6
  % Recurrence Free by Day 56: number analyzed (Participants) | 23 | 14
  % Recurrence Free by Day 56 | 55.5 | 42.2

6. Secondary Outcome: Time to CDAD Recurrence After Completion of the Assigned Study Treatment for Group C vs. Group B (ITT)
Description: as for outcome 5
Time Frame: 8-weeks
Population: ITT
Measure: Number; unit: percentage of participants
Groups:
- Group C: One enemas of RBX2660 (microbiota suspension) and one enema of Placebo administered 7 days apart
  RBX2660 (microbiota suspension): A suspension of intestinal microbes Placebo: A suspension of saline and cryoprotectant
Arm/Group | Group C | Group B
Number analyzed (Participants) | 44 | 44
percentage of participants
  % Recurrence Free by 2nd Enema | 95.5 | 100
  % Recurrence Free by Day 7: number analyzed (Participants) | 37 | 35
  % Recurrence Free by Day 7 | 76.9 | 77.3
  % Recurrence Free by Day 14: number analyzed (Participants) | 31 | 30
  % Recurrence Free by Day 14 | 69.9 | 63.6
  % Recurrence Free by Day 21: number analyzed (Participants) | 28 | 27
  % Recurrence Free by Day 21 | 62.9 | 61.4
  % Recurrence Free by Day 28: number analyzed (Participants) | 27 | 25
  % Recurrence Free by Day 28 | 62.9 | 56.8
  % Recurrence Free by Day 35: number analyzed (Participants) | 26 | 23
  % Recurrence Free by Day 35 | 60.6 | 52.3
  % Recurrence Free by Day 42: number analyzed (Participants) | 25 | 22
  % Recurrence Free by Day 42 | 55.9 | 50.0
  % Recurrence Free by Day 49: number analyzed (Participants) | 23 | 21
  % Recurrence Free by Day 49 | 55.9 | 47.6
  % Recurrence Free by Day 56: number analyzed (Participants) | 20 | 14
  % Recurrence Free by Day 56 | 55.9 | 42.2

7. Secondary Outcome: Time to CDAD Recurrence After Completion of the Assigned Study Treatment for Group A vs. Group C (ITT)
Description: as for outcome 5
Time Frame: 8-weeks
Population: ITT
Measure: Number; unit: percentage of participants
Groups:
- Group C: One enema of RBX2660 (microbiota suspension) and one enema of Placebo administered 7 days apart
  RBX2660 (microbiota suspension): A suspension of intestinal microbes Placebo: A suspension of saline and cryoprotectant
Arm/Group | Group A | Group C
Number analyzed (Participants) | 45 | 44
percentage of participants
  % Recurrence Free by 2nd Enema | 91.1 | 95.5
  % Recurrence Free by Day 7: number analyzed (Participants) | 35 | 37
  % Recurrence Free by Day 7 | 73.3 | 76.9
  % Recurrence Free by Day 14: number analyzed (Participants) | 30 | 31
  % Recurrence Free by Day 14 | 66.7 | 69.9
  % Recurrence Free by Day 21: number analyzed (Participants) | 27 | 28
  % Recurrence Free by Day 21 | 60.0 | 62.9
  % Recurrence Free by Day 28: number analyzed (Participants) | 27 | 27
  % Recurrence Free by Day 28 | 60.0 | 62.9
  % Recurrence Free by Day 35: number analyzed (Participants) | 27 | 26
  % Recurrence Free by Day 35 | 57.8 | 60.6
  % Recurrence Free by Day 42: number analyzed (Participants) | 26 | 25
  % Recurrence Free by Day 42 | 57.8 | 55.9
  % Recurrence Free by Day 49: number analyzed (Participants) | 24 | 23
  % Recurrence Free by Day 49 | 55.5 | 55.9
  % Recurrence Free by Day 56: number analyzed (Participants) | 23 | 20
  % Recurrence Free by Day 56 | 55.5 | 55.9

ADVERSE EVENTS:
Time Frame: 24 months
Description: Data reported here is from the Safety Population, defined as randomized subjects who received any study treatment. The adverse events presented were captured during the double-blind portion of the study. Subjects who were deemed treatment failures had an opportunity to access additional RBX2660 open-label doses, and any open-label treatment emergent adverse events in the open-label period are not presented here.
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 7/42 | 2/44 | 6/42
Serious Adverse Events (participants affected / at risk) | 18/42 | 8/44 | 12/42
Other Adverse Events (participants affected / at risk) | 24/42 | 19/44 | 20/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=42) | Group B (N=44) | Group C (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcimoa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Malocclusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (3) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=42) | Group B (N=44) | Group C (N=42)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 3 (3) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 10 (13) | 8 (10) | 8 (9)
Anorectal discomfort (Gastrointestinal disorders) | 3 (4) | 3 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 17 (27) | 7 (10) | 5 (7)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (8) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (9) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 4 (4) | 2 (2) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Chills (General disorders) | 2 (5) | 4 (5) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 5 (11) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No